CLINICAL TRIAL: NCT03110692
Title: Health System Initiative to Reduce Unnecessary Daily X-Ray Image Guidance During Palliative Radiation Treatment
Brief Title: Default Options to Reduce Unnecessary Daily Imaging During Palliative Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 826810
Record Dates: First submitted 2017-03-29; First posted 2017-04-12 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual practice (control) (No Intervention): The usual practice group will rollover to the intervention arm after 3 months.
- Intervention (Experimental): Default initiation: Introduce a default prescription template in the palliative setting in order to reduce unnecessary daily image guided radiation.
  Interventions: Behavioral: Default initiation

INTERVENTIONS:
Behavioral: Default initiation — A default prescription template will be introduced in the palliative setting in order to reduce unnecessary daily image guided radiation.
  Arms: Intervention

SUMMARY:
The goal of this study is to reduce preference sensitive, unnecessary daily imaging during radiation treatment in which a pre-planned quality improvement default option for radiation treatment prescriptions will be introduced throughout the network of Penn Radiation Oncology.

DETAILED DESCRIPTION:
The goal of this study is to reduce preference sensitive, unnecessary daily imaging during radiation treatment in which a pre-planned quality improvement default option for radiation treatment prescriptions will be introduced throughout the network of Penn Radiation Oncology. This study is a prospectively designed, observational trial with two comparison groups: (1) a usual practice group (control group) and (2) a default radiation treatment prescription group (intervention group), in which the usual practice group will subsequently rollover from control to intervention so that all sites and physicians in the practice network of Penn Radiation Oncology are exposed to intervention. The purpose of this study is to reduce preference sensitive, unnecessary daily imaging during radiation treatment with the implementation of a quality improvement initiative within 5 sites of Penn Radiation Oncology. We aim to leverage the introduction of a default prescription option to reduce the use of daily imaging in palliative intent cases where it has limited clinical benefit and adds to cost burden. Our objective is to encourage more patient-centric clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Radiation treatment courses with palliative intent
* Palliative treatment of bone, soft tissue, and intracranial metastases
* Photon radiation with 3D conformal therapy (3DCRT) only

Exclusion Criteria:

* Use of intensity modulated radiation (IMRT) or stereotactic body radiation (SBRT) as radiation treatment modality
* Retreatment to same site
* Proton radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1188 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Bekelman, MD, Principal Investigator — University of Pennsylvania; Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma S, Guttmann D, Small DS, Rareshide CAL, Jones J, Patel MS, Bekelman JE. Effect of Introducing a Default Order in the Electronic Medical Record on Unnecessary Daily Imaging During Palliative Radiotherapy for Adults With Cancer: A Stepped-Wedge Cluster Randomized Clinical Trial. JAMA Oncol. 2019 Aug 1;5(8):1220-1222. doi: 10.1001/jamaoncol.2019.1432. PMID 31246224

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Practice (Control): The usual practice group will rollover to the intervention arm 3 months after the start of the default intervention group in Feb. 2017
- Intervention: Default initiation: Introduce a default prescription template in the palliative setting in order to reduce unnecessary daily image guided radiation.
  Default initiation: A default prescription template will be introduced in the palliative setting in order to reduce unnecessary daily image guided radiation.
  To start in Feb 2017 and continue in the intervention through Feb 2018
Period: Overall Study
Arm/Group | Usual Practice (Control) | Intervention
Started | 679 | 509
Completed | 679 | 509
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Practice (Control): The usual practice group will rollover to the intervention arm after 3 months following the start of the default intervention in Feb 2017.
- Total: Total of all reporting groups
Arm/Group | Usual Practice (Control) | Intervention | Total
Number analyzed (Participants) | 679 | 509 | 1188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 341 | 259 | 600
  >=65 years | 338 | 250 | 588
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 347 | 268 | 615
  Male | 332 | 241 | 573
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White non-hispanic | 470 | 333 | 803
  Race/Ethnicity: Black non-hispanic | 147 | 114 | 261
  Race/Ethnicity: Other | 41 | 37 | 78
  Race/Ethnicity: Missing | 21 | 25 | 46
ECOG Performance Status [Number; unit: participants] — The ECOG (Eastern Cooperative Oncology Group) Performance Status is used to classify a patient according to their functional status. It assesses how the disease affects the daily living abilities of the patient, and to help determine treatment and prognosis.
  Scale Ranking 0- Fully active, able to carry on all pre-disease performance without restriction
  1 2 3- 4-Completely disabled, cannot carry on any selfcare, totally confined to bed or chair
  participants
    0 | 92 | 66 | 158
    1 | 200 | 145 | 345
    2 | 206 | 133 | 339
    3 | 151 | 121 | 272
    4 | 27 | 26 | 53
    Missing | 3 | 18 | 21
Insurance [Count of Participants; unit: Participants]
  Medicaid | 46 | 54 | 100
  Medicare | 337 | 226 | 563
  Commercial | 296 | 229 | 525
Target Type [Count of Participants; unit: Participants]
  Bone | 345 | 275 | 620
  Brain | 104 | 82 | 186
  Soft Tissue | 133 | 103 | 236
  Multiple Sites | 97 | 49 | 146
Prior Radiation [Count of Participants; unit: Participants] | 381 | 268 | 649
Number of Patients Receiving Fractions [Count of Participants; unit: Participants] — The measure shows the proportion of patients that received X number of fractions per course
  Participants
    2-5 total fractions per course | 156 | 162 | 318
    6-10 total fractions per course | 403 | 277 | 680
    11-15 total fractions per course | 104 | 51 | 155
    15+ total fractions per course | 16 | 19 | 35
Number of patients receiving dose per fraction [Count of Participants; unit: Participants] — The total radiation dose is divided up into several fractions. Each fraction contains a small amount of radiation that gradually accumulates to form the total dose. The measure displayed shows the proportion of patients that received the dose per fraction.
  Participants
    Less than or equal to 200 doses per fraction | 26 | 38 | 64
    201-300 doses per fraction | 509 | 308 | 817
    301-400 doses per fraction | 137 | 154 | 291
    Greater than 400 doses per fraction | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Receiving Daily Imaging
Description: Radiology tests including x-rays and CT scans
Time Frame: 3 months post arm crossover
Measure: Count of Participants; unit: Participants
Groups:
- Usual Practice (Control): The usual practice group will rollover to the intervention arm after 3 months from start of the default intervention in Feb 2017.
Arm/Group | Usual Practice (Control) | Intervention
Number analyzed (Participants) | 679 | 509
Participants | 679 | 509

ADVERSE EVENTS:
Time Frame: Through study completion (1 year from study start)
Arm/Group | Usual Practice (Control) | Intervention
All-Cause Mortality (participants affected / at risk) | 0/679 | 0/509
Serious Adverse Events (participants affected / at risk) | 0/679 | 0/509
Other Adverse Events (participants affected / at risk) | 0/679 | 0/509

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT03110692/SAP_000.pdf
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03110692/Prot_001.pdf